CLINICAL TRIAL: NCT04738357
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of HSK21542 Injection for Postoperative Analgesia of Subjects Undergoing Elective Laparoscopic Surgery Under General Anesthesia
Brief Title: A Clinical Study to Evaluate Efficacy and Safety of HSK21542 for Postoperative Analgesia of Subjects Undergoing Elective Laparoscopic Surgery Under General Anesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK21542-301
Record Dates: First submitted 2021-01-31; First posted 2021-02-04 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-05

CONDITIONS: Postoperative Analgesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK21542 (Experimental)
  Interventions: Drug: HSK21542
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK21542 — HSK21542：1 µg/kg
  Arms: HSK21542
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
This study is a multi-center, randomized, double-blind, placebo-controlled study. A total of 276 subjects undergoing elective laparoscopic surgery under general anesthesia are planned to be enrolled and randomized into 2 groups, i.e., the HSK21542 group (138 subjects) and the placebo group (138 subjects).

ELIGIBILITY:
Inclusion Criteria:

1. 18 ≤ age ≤ 70 years old, with no gender requirement;
2. American Society of Anesthesiologists (ASA) Class I-II;
3. BMI ≥ 18 kg/m2 and ≤ 40 kg/m2;
4. Subjects undergoing elective laparoscopic surgery under general anesthesia with an expected surgery duration of 1-5 h (inclusive);
5. Agree to participate in this trial and voluntarily sign the informed consent form;

Exclusion Criteria:

1. With a history of allergy to opioids, such as urticaria, or allergic to intraoperative anesthetics as prescribed in the protocol;
2. Patients with history or evidence of any of the following diseases prior to screening:

   1. History of cardiovascular diseases: uncontrolled hypertension (systolic blood pressure [SBP] ≥ 170 mmHg and/or diastolic blood pressure [DBP] ≥ 105 mmHg without treatment, or SBP > 160 mmHg and/or DBP > 100 mmHg despite antihypertensive treatment), aneurysm, severe arrhythmia, heart failure, Adams-stokes syndrome, New York Heart Association (NYHA) Class ≥ III, severe superior vena cava syndrome, pericardial effusion, acute myocardial ischemia, unstable angina, myocardial infarction within 6 months before screening, history of tachycardia/bradycardia requiring medical treatment, II-III degree atrioventricular block (excluding patients with pacemakers);
   2. History of respiratory system disorders: severe chronic obstructive pulmonary disease, acute exacerbation of chronic obstructive pulmonary disease, severe airway stenosis, throat mass, history of tracheoesophageal fistula or airway tear, severe respiratory infection within 2 weeks prior to screening;
   3. History of neurological and psychiatric disorders: craniocerebral injury, convulsions, intracranial hypertension, cerebral aneurysms, history of cerebrovascular accidents; schizophrenia, mania, insanity, long-term use of psychotropic drugs, and history of cognitive dysfunction; history of depression, anxiety, and epilepsy, etc.;
   4. Have undergone any major surgery within 3 months prior to screening, which may affect postoperative pain assessment as judged by the investigator;
3. In receipt of any one of the following medications or treatments at screening:

   1. A time between the last use of opioid and non-opioid (such as paracetamol, aspirin [daily dose > 100 mg], indometacin, diclofenac, parecoxib sodium, and other non-steroidal anti-inflammatory drugs) analgesics and randomization of shorter than 5 half-lives of the drug or the duration of response (whichever is longer);
   2. Longer than 10 days of continuous use of opioid analgesics for any reason within 3 months prior to screening;
   3. Use of drugs with unknown half-life that affect the analgesic effect within 14 days before randomization, or the last use of drugs that affect the analgesic effect is within 5 half-lives (as per the packaging insert of the drug) apart from randomization, such drugs include but are not limited to: sedative-hypnotics (benzodiazepines [triazolam, diazepam, midazolam, etc.], non-benzodiazepines [zolpidem, zopiclone, zaleplon, etc.]), sedative anesthetics (sevoflurane, anesthetic ether, nitrous oxide, thiopental sodium, ketamine, etomidate, etc.), glucocorticoids (dexamethasone hydrochloride, methylprednisolone, etc.), antiepileptics (carbamazepine, sodium valproate, etc.), anxiolytics (chlordiazepoxide, diazepam, etc.), antidepressants (imipramine, amitriptyline, etc.), and Chinese herbal medicines or Chinese patent medicines with analgesic and sedative effects;
   4. Expected to receive any anti-tumor drug or therapy from 14 days prior to randomization to the end of the follow-up period, including but not limited to chemotherapy drugs, targeted drugs, and Chinese herbal medicines;
   5. A time between randomization and the last use of diuretics and compound drugs containing diuretics of shorter than 5 half-lives of the drug or the duration of response (whichever is longer);
4. The laboratory parameters measured at screening period reach one of the following criteria:

   1. WBC < 3.0 × 109/L;
   2. Platelet count < 80 × 109/L;
   3. Hemoglobin < 70 g/L;
   4. Prothrombin time > 1.5 × ULN;
   5. Activated partial thromboplastin time > 1.5 × ULN;
   6. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 2 × ULN;
   7. Total bilirubin > 1.5 × ULN;
   8. Blood creatinine > 1.5 × ULN;
   9. Fasting blood glucose ≥ 11.1 mmol/L;
5. Positive for hepatitis C antibody (HCVAb), syphilis antibody, or human immunodeficiency virus (HIV) antibody at screening;
6. History of medication or drug abuse and/or alcohol abuse within 3 months prior to screening (alcohol abuse is defined as an average of > 2 units of alcohol consumed per day [1 unit = 360 mL of beer with 5% alcohol, 45 mL of liquor with 40% alcohol, or 150 mL of wine]);
7. History of blood donation or blood loss of ≥ 400 mL within 3 months prior to screening;
8. Have participated in other clinical trials within 3 months prior to screening (defined as having received investigational product or placebo);
9. Pregnant or breastfeeding females; women of child-bearing potential or men who are unwilling to use contraception during the trial; or subjects who are planning pregnancy within 3 months after the completion of the trial (including male subjects);
10. Subject judged by the investigator to have any other factors unsuitable for involvement in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Sum of Pain Intensity Differences (SPID) | Frome administration until 24 hours after administration
  The time-weighted SPID at rest within 0-24 h after the first postoperative administration in each group

SECONDARY OUTCOMES:
Sum of Pain Intensity Differences (SPID) | Frome administration until 12 hours after administration
  The time-weighted SPID at rest within 0-12 h after the first postoperative administration in each group
Use of remedial analgesics | Frome administration until 24 hours after administration
  Cumulative used amount of remedial analgesics (morphine injection, mg) within 0-12 h or 0-24 h after the first postoperative administration in each group, percentage of subjects not using remedial analgesics, and start time of remedial analgesic use
Pain Intensity Differences（PID） | Frome administration until 24 hours after administration
  The PID at rest at each scoring time point after the first postoperative administration in each group
The proportion of subjects with a NRS of ≤ 3 | Frome administration until 24 hours after administration
  The ratio of subjects with NRS score ≤ 3 at 12 h or 24 h after the first postoperative administration in each group
Duration of analgesia | Frome administration until 24 hours after administration
  The duration of analgesia after the first postoperative administration in each group
Satisfaction scores on postoperative analgesia | Frome administration until 24 hours after administration
  Subject satisfaction score and investigator satisfaction score on postoperative analgesia at 24 h after the first postoperative administration in each group
The incidence and severity of AEs | from signing the informed consent form to the follow-up period (D8 ± 1 postoperative).
  Adverse event/serious adverse event
Cumulative used amount and ratio of antiemetics | Frome administration until 24 hours after administration
  Cumulative used amount and ratio of antiemetics within 0-24 h after the first postoperative administration in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, China

REFERENCES:
- [Derived] Zhong Y, Xu Y, Lei Q, Yang M, Wang S, Hu X, Xie H, Li Y, Qin Z, Gu Z, Zhang J, Wang Y, Wu J, Wang H, Ming Y, Xia Z, Zhai H, Jiang K, Zhang P, Wang Z, Wang L, Li L, Cheng Z, Jiang H, Wang G, Chen J, Zhao Z, Chen X, Yan M. HSK21542 in patients with postoperative pain: two phase 3, multicentre, double-blind, randomized, controlled trials. Nat Commun. 2025 May 24;16(1):4830. doi: 10.1038/s41467-025-60013-y. PMID 40413233